CLINICAL TRIAL: NCT02275299
Title: A Randomized, Double-blind Study to Evaluate the Efficacy and Safety of Iguratimod or Leflunomide in Combination With Methotrexate in Patients With Active Rheumatoid Arthritis
Brief Title: Study of Iguratimod Plus Methotrexate Compared to Leflunomid Plus Methotrexate in Patients With Rheumatoid Arthritis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Tranmod
Record Dates: First submitted 2014-10-23; First posted 2014-10-27 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2014-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — iguratimod; Leflunomide; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Iguratimod and MTX combination (Experimental): Drug:Iguratimod 25 mg/tablet, taken orally, 2 tablets/day (bid) Drug:MTX 2.5 mg/tablet, taken orally once a week, 4 tablets/week
  Interventions: Drug: Iguratimod; Drug: Methotrexate
- Leflunomide and MTX combination (Active Comparator): Drug: Leflunomide 10 mg/tablet, taken orally, 2 tablets/day (bid) Drug: Methotrexate 2.5 mg/tablet, taken orally once a week, 4 tablets/week
  Interventions: Drug: Leflunomide; Drug: Methotrexate

INTERVENTIONS:
Drug: Iguratimod — Iguratimod 25 mg/tablet, taken orally, 2 tablets/day (bid),52 weeks
  Other Names: Iremod
  Arms: Iguratimod and MTX combination
Drug: Leflunomide — Leflunomide 10 mg/tablet, taken orally, 2 tablets/day (bid),52 weeks
  Arms: Leflunomide and MTX combination
Drug: Methotrexate — Methotrexate 2.5 mg/tablet, taken orally once a week, 4 tablets/week,52 weeks

SUMMARY:
This study is intended to evaluate the efficacy and safety of Iguratimod Plus Methotrexate Compared to Leflunomid Plus Methotrexate in patients with active Rheumatoid Arthritis (RA).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a diagnosis of RA according to the diagnostic criteria of the American College of Rheumatology (ACR) (revised in 1987)
* Rheumatoid Arthritis for more than 3 months from the time of the initial diagnosis
* Functional Class II-III
* Subjects have active RA at the time of screening
* Subjects with inadequate response to biologics should have a washout period before the initiation of study. For etanercept, washout period should be 2-week, and 8-week for infliximab and adalimumab.
* For firstly diagnostic RA patients, the disease activity should be moderate to severe, with DAS28>3.2
* Must have at least 4 tender joints (66 join count) and 8 swollen joints( 68 join count) at screening and baseline
* Has a C-reactive protein ≥ 10 mg/L(or 1.0 mg/dL) OR Erythrocyte Sedimentation Rate (ESR) ≥ 28 mm/hr
* Must have a negative Pregnancy test and use adequate method of contraception throughout the trial
* Written informed consent

Exclusion Criteria:

* Preceding treatment with DMARDs, immunosuppressants (cyclophosphamide, cyclosporine, azathioprine, etc.), or Tripterygium within 4 weeks prior to study entry
* Subjects have been treated with iguratimod or leflunomide combined with MTX before screening.
* Subjects combined with other autoimmune disease, such as systemic lupus erythematosus (SLE), mixed connective tissue disease (MCTD), scleriasis and polymyositis, except for Sjögren syndrome.
* Chest x-ray abnormalities, such as tuberculosis, interstitial pulmonary fibrosis, etc.
* ALT >1.5×ULN, AST >1.5×ULN, Cr >135umol/L, total bilirubin>1.5×ULN
* WBC<4×109/L，HGB<85g/L，PLT<100×109/L
* Subjects with serious cardiovascular, renal, hematologic, endocrine diseases or malignant
* Women of Pregnant or breastfeeding, and male or female with recent plan to conception
* Subjects with immunodeficiency, uncontrolled infection and active gastrointestinal disease
* Allergic to any of the study drugs
* History of alcoholism
* Subjects with mental illness
* Subjects receiving live vaccines recently
* Subjects participating in other clinical study within 3 months prior to study entry

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2013-09; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with ACR 20 response and Change in Disease Activity as measured by the DAS28 | week 52

SECONDARY OUTCOMES:
Change from baseline in modified Total Sharp Score (mTSS) | week 52
Percentage of patients with ACR 50 response and ACR70 response | week 24,week 52
Change from baseline in number of swollen and tender joins, Erythrocyte sedimentation rate (ESR) ,C-reactive protein (CRP),anti-citrullinated-protein antibody (ACPA) and heumatoid factor(RF) | week 24, week 52
Time to achieve the ACR20, ACR50 and ACR70 | week 12, week 24, week 40, week 52
Percentage of patients with Simplified Disease Activity Index (SDAI) ≤ 3.3 and change from baseline in Health Assessment Questionnaire (HAQ) | week 12, week 24, week 40, week 52
Incidence of adverse events | up to 52 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China